CLINICAL TRIAL: NCT06471179
Title: Functional Magnetic Resonance Imaging Study of Schizophrenic Patients and Its Correlation With Cognitive Impairments
Brief Title: Functional Magnetic Resonance Imaging Study in Schizophrenia Patients and Correlation With Cognitive Impairments
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, waleed ashraf hamdy ahmed, Principal investigator, Assiut University
Other Study IDs: fMRI in schizophrenia
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Cognitive Impairment
Keywords: Functional MRI; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A Patients: Schizophrenic patients according to diagnostic criteria
  Interventions: Device: Functional MRI
- group B Control: healthy subjects not suffering from any Psychiatric illness
  Interventions: Device: Functional MRI

INTERVENTIONS:
Device: Functional MRI — Functional Magnetic Resonance Imaging during rest for minutes and analysis of data obtained from resting fMRI

SUMMARY:
1. Comparison of functional activity at different brain areas related to different cognitive domains e.g. Memory, visuospatial abilities, executive functions, attention, concentration, language, orientation in schizophrenia to healthy subjects.
2. Correlation with resting functional activity at brain areas with clinical deterioration in cognitive functions.

DETAILED DESCRIPTION:
Schizophrenia represents a multifaceted clinical challenge. Patients' outcome is still highly heterogeneous and poor. Cognitive impairment, a central feature of the illness is present in over 80% of patients with schizophrenia, is a main functional disability. Currently available antipsychotics have only limited effects on cognition and side effects may even aggravate some deficits. So far, pharmacological options for cognitive deficits in schizophrenia are unsatisfactory due to either limited efficacy or tolerability concerns. Understanding the quality, quantity of brain changes could cover patterns of potential therapeutic relevance, guiding treatments. Understanding the pathophysiology of impaired cognition in schizophrenia and developing effective treatment for cognitive symptoms are major unmet challenges for contemporary biomedical research. Briefly, deficits in speed of processing have been correlated with a reduced temporal lobe volume and increased ventricular size. Attention impairments were correlated with structural alterations within the frontal and temporal lobes and with widespread reduced volume of subcortical regions . Decreased working memory was correlated with reduced frontal and temporal lobe volumes and cortical thickness while language and memory deficits were correlated with hippocampal volume loss. Impaired visuspatial and memory correlated with hippocampal volume loss. Deficits in reasoning and problem solving, including higher-order executive functions, were also associated with a reduced the dorsolateral prefrontal cortex volume. Among different neuroimaging modalities, functional magnetic resonance imaging (fMRI) predominates in system-level connectomic studies. Particularly, the task-free version-known as resting fMRI-is better tolerated by clinical populations, and circumvents the need for stringent subject compliance. Today, fMRI features are being rigorously examined to identify potential biomarkers for diagnosis and prognosis of different brain disorders

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis according to Diagnostic and statistical manual of mental of mental disorders -5 (DSM-5) and confirmed by the Structured Clinical Interview for DSM-5 (SCID -I)

Exclusion Criteria:

* History of head injury.
* History of intellectual disability or neurological diseases e.g. cerebrovascular stroke, dementia Parkinsonism, etc.
* History of alcohol and/or substance abuse in the previous six months.
* Inability to provide informed consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: twenty subjects will be chosen from psychiatric inpatient unit from assiut university hospitals diagnosed with schizophrenia and 20 subjects as control to be investigated for affection of brain activity in case of schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
functional Magnetic Resonance Imaging | baseline
  different regional brain activity among schizophrenic and healthy subjects and correlation with cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Wageeh A Hassan, MD, Study Chair — Assiut University; Hossam E Khalifa, Study Director — Assiut University